CLINICAL TRIAL: NCT04018092
Title: Revitalizing Cognition in Older Adults at Risk for Alzheimer's Disease With Near-Infrared Photobiomodulation
Brief Title: The Revitalize Study in Older Adults at Risk for Alzheimer's Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of Arizona (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB201901780 -N; R01AG064587 (NIH); F31AG071264 (NIH)
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-06

CONDITIONS: Cognitive Aging; Alzheimer Disease, Protection Against
MeSH Terms: conditions — Alzheimer Disease | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Randomized, sham-controlled: Participants who meet eligibility criteria will be randomized to the Active or Sham condition. The study biostatistician will randomize participants using a 1:1 allocation scheme with stratification based on age, education, and sex. When a new participant arrives, she/he will be randomized to Active or Sham groups depending on covariate characteristics (age, education, sex) and the cumulative distribution of assignments regarding these variables at that point.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Use of a sham-controlled approach provides stringent experimental control, enabling the investigators to control for placebo/expectations, behavioral activation (engaging in study procedures) and practice effects related to repeated administration of the same cognitive tasks.
  The MedX and Vielight devices used for delivery of active and sham NIR stimulation are identical in all respects regarding design, warmth and operation, except that no stimulation is delivered by the sham devices. Because NIR light is invisible, participants will not be able to discern if receiving active or sham stimulation. The participants, interventionists, and outcome assessors will be blinded to the participants' intervention status: Active vs Sham. At completion of the study, all participants will receive a Placebo Control Questionnaire that asks questions pertaining to what group the participant had been assigned. This data will be examined to determine the effectiveness of blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active NIR-PBM (Experimental): This condition involves baseline testing, 12 weeks of Near Infrared-Photobiomodulation (NIR-PBM), and post-intervention testing. Cognitive and neuroimaging outcomes are obtained before and after the intervention. The intervention consists of a) 16 laboratory sessions of NIR-PBM given 3 times/week for 2 weeks and then once weekly for 10 weeks and b) 44 home sessions of stimulation delivered intranasally. During each lab session, NIR light is delivered via placement of six MedX LED superluminous diode clusters over the scalp for a total of 40 minutes. Concurrently, two 810 Vielight intranasal devices are placed in each nostril for 25 min of total dose per nostril. During lab sessions, participants sit in front of a monitor and view nature documentaries (BBC Life series). This is done to standardize behavior during the intervention sessions. For home sessions, participants use a standalone 810 intranasal device only on weekdays when not completing a lab session.
  Interventions: Device: Active NIR-PBM
- Sham NIR-PBM (Sham Comparator): Participants randomized to the Sham control group will undergo identical procedures as the Active group. The only difference is that the "sham" NIR devices are modified not to deliver stimulation. Because NIR is invisible, participants are unable to detect whether NIR is being delivered.
  Interventions: Device: Sham NIR-PBM

INTERVENTIONS:
Device: Active NIR-PBM — Near infrared light was delivered to the head using two MedX Rehab Console systems (MedX Health, 1116). Each MedX console included a control unit and 3 superluminous light emitting diode (LED) clusters. Each LED cluster (3MedX MCT502) consisted of 52 near infrared diodes and 9 visible red diodes. The 9 red diodes were deactivated. The energy delivered by each cluster was 1 joule [J]/cm2 in 45 sec at treatment wavelength of 870 nm per each 20 min. The LED cluster has an irradiance of 22.2 mW/cm2, treats an area of 22.48 cm2, with an energy density of 26.64/cm2 per cluster (total energy of 599J/cluster). During each session, the 6 clusters were arrayed on the scalp in 2 configurations, 20 minutes per array. Each configuration targeted 6 transcranial sites, guided by the 10-20 system, for a total of 12 sites during the 40-min session. Total energy delivered was 599J/cluster X 12 sites = 7188J. Intranasal stimulation was delivered using..
  Other Names: Transcranial Near Infrared Stimulation; Photobiomodulation
  Arms: Active NIR-PBM
Device: Sham NIR-PBM — The MedX sham and Vielight interventions device are identical in all respects to the active device, except that the MedX console and diode clusters were modified to NOT deliver NIR light when turned on. The sham MedX devices were modified to deliver 'warmth', similar to that of the active devices. As with the active condition, a total of six sham interventions were given over a 12-week period, following the identical procedures described in the active condition
  Arms: Sham NIR-PBM

SUMMARY:
The goal of this multi-site double blinded randomized sham-controlled Phase II clinical trial is to test a novel, relatively low cost, low risk, and potentially high impact therapeutic intervention in older adults who are at increased risk for Alzheimer's disease. The intervention involves transcranial and intranasal delivery of near infrared (NIR) light via light emitting diodes, aka photobiomodulation (PBM). The overall hypothesis, based on animal and pilot studies, is that exposure to NIR stimulation will have beneficial effects on brain health via influence on mitochondrial function as measured by changes in 31Phosphorous (31P) MRS-based markers of ATP, neural network changes in functional connectivity (rs-fMRI), and improved cognitive performance. To test this hypothesis, 168 older adults with subjective cognitive complaints, and a first-degree family history of Alzheimer's disease will be randomized to sham or real treatment groups. Neuroimaging and cognitive outcome measures will be obtained, before and after a 12-week intervention involving transcranial and intranasal NIR-PBM. The intervention protocol will involve "lab" and "home" sessions, and a 3 month post-intervention follow-up. This trial will determine: 1) whether NIR stimulation, relative to sham, improves performance on memory and executive tasks sensitive to hippocampal and frontal brain function in older adults with increased risk for Alzheimer's disease; 2) whether NIR stimulation, relative to sham, enhances brain function and connectivity measured by changes in MRS phosphorous ATP and resting state functional connectivity; and 3) how differences in demographic, neuroimaging, and Alzheimer-related risk factors influence the brain response to NIR stimulation versus sham in older adults with increased risk for Alzheimer's disease. Results will provide key insights into whether this novel NIR intervention can enhance cognition in older adults with increased risk for Alzheimer's disease and will provide the necessary data for a future Phase III randomized clinical trial.

DETAILED DESCRIPTION:
This multi-site randomized sham-controlled trial proposes to test a novel, non-invasive, low risk and low-cost brain stimulation approach for enhancing cognition and brain health in cognitively normal older adults who are at increased risk for Alzheimer's disease. The intervention involves transcranial and intranasal delivery of near-infrared light (NIR; 808-904 nm) via light emitting diodes placed on the scalp or intranasally using a dosing that resulted in positive effects in our pilot studies. We plan to test the hypothesis that targeted NIR stimulation will have positive effects on brain health via influence on mitochondrial function as measured by changes in Magnetic Resonance Spectroscopy (MRS)-based markers of adenosine triphosphate (ATP), neural network changes as indexed by changes in functional connectivity based on resting state-fMRI (rs-fMRI), and improved cognitive performance. We plan to randomize 168 older adults, ages 65-89 years, to Active or Sham intervention conditions. To be included, participants must have subjective cognitive complaints, based on an index of Subjective Cognitive Impairment (SCI), and a family history of Alzheimer's disease in a first degree relative. Performance on standardized neuropsychological measures must be unimpaired psychometrically. The intervention itself will last for 12 weeks and include lab sessions (16 total) and daily at home sessions. In the lab, both transcranial and intranasal delivery of NIR light will be delivered using Medx and Vielight stimulation technologies, whereas the daily at home sessions will involve intranasal stimulation only. The sham and active conditions are identical in all respects except that sham devices will not deliver NIR stimulation. The primary outcome is an episodic memory measure involving spatial navigation that is linked to hippocampal function, sensitive to mild cognitive impairment (MCI) and Alzheimer's disease, and an analogue to the Morris Water maze. Secondary outcomes include executive function tasks and neuroimaging indicators of ATP function (31-P MRS) and connectivity changes based on resting state-fMRI. Exploratory outcomes include 'traditional' neuropsychological measures that are used clinically, along with measures and indices (e.g., apolipoprotein E [APOE-4] status) that might potentially mediate or moderate study outcome. Assessments will occur at baseline (Month 1), after 12 weeks of intervention (Month 4), and 3-month post intervention (Month 7). Imaging outcomes will be assessed only at baseline and at Month 4. Our primary aim is focused on cognition and will test whether NIR intervention, relative to sham, will produce pre-post improvement on tasks of recent memory (primary outcome) and executive function in older adults who are at increased risk for Alzheimer's disease. Our secondary aim is focused on neuroimaging and will test whether NIR intervention, relative to sham, will increase functional connectivity as indexed by resting state fMRI (secondary outcome) and enhance brain markers of MRS-ATP (secondary outcome). The 3rd aim is exploratory and will evaluate how baseline demographic, genetic, neuroimaging and other factors influence individual differences in cognitive outcome for NIR intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-89 years, at least 8th grade education, community dwelling
* Subjective report of cognitive complaints with scores >16 on the Cognitive Change Index (CCI-20)
* No evidence of dementia or mild cognitive impairment based on cognitive screening (i.e., Montreal Cognitive Assessment (MoCA) score within normal limits for age, education and sex using the National Alzheimer's Coordinating Center (NACC) Uniform Data Set (UDS) norms.
* No psychometric evidence of cognitive impairment based on performance on the Neuropsychological Battery from the NACC Unified Data Set, version 3. Scores on these measures cannot be lower than 5th percentile below normative values based on age, education, and gender.
* Reading at > 8th grade level based on the reading subtest of the Wide Range Achievement Test- IV.
* Global Clinic Dementia Rating (CDR) score must be 0
* Family history of dementia/probable Alzheimer's disease in first degree relative (parents, children, siblings)
* Willingness to be randomized to Sham or Active Intervention
* Can devote 12 weeks to the intervention with additional time for pre and post testing
* Normal functional behavior in terms of daily activities, based on the Functional Activities Scale
* Able to perform cognitive and emotion measures on a computer
* In line with recommendations of the Subjective Cognitive Decline (SCD) task force an informant must be available for two reasons: a) to provide information about the participant's complaints using the informant version of the CCI-20, and b) to corroborate normal IADL's on the Functional Activity Questionnaire.

Exclusion Criteria:

* Sensory loss (vision, hearing) or motor deficits that would preclude participation in the experimental tasks or neuropsychological assessment
* English as a second language
* Inability to undergo brain imaging due to claustrophobia or implants such as pacemakers, heart valves, brain aneurysm clips, orthodontics, non-removable body jewelry, or shrapnel containing ferromagnetic metal
* Previous major strokes or other known significant brain abnormalities or diseases affecting the brain and/or cognition (e.g.,Parkinson disease, multiple sclerosis, seizure disorder, brain surgery, moderate traumatic brain injury (TB)I, Rapid Eye Movement (REM) Behavior Sleep Disorder, untreated sleep apnea, etc.)
* Unstable and uncontrolled medical conditions (metastatic cancer, HIV, moderate-severe kidney disease, uncontrolled diabetes, uncontrolled hypertension, severe cardiac disease, etc.). No current cancer diagnosis.
* Current or past history of major psychiatric disturbance including schizophrenia, or active psychosis, bipolar disorder, current major depressive episode, current alcohol or substance abuse or history thereof within the past six months.
* Use of antipsychotics, sedatives, or other medications with significant anticholinergic properties (due to potential influence on memory)
* Use of prescribed 'memory enhancing' medications such as Aricept or Namenda
* Use of photo-sensitive medications such as steroids or retin-A within 15 days of the study intervention.
* Previous participation in a cognitive training study within the last 6 months or current involvement in another study involving cognitive, physical or other intervention at the time of participation

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 168 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Bowers, Ph.D, Principal Investigator — University of Florida; Steve DeKosky, M.D., Principal Investigator — University of Florida; Gene Alexander, Ph.D., Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - University of Florida McKnight Brain Institute, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment began August 12, 2020 and ended in 2024, across the University of Florida and University of Arizona sites.
Pre-assignment Details: No participants were randomized until they met inclusion-exclusion criteria and completed baseline assessments. A total of 345 participants were screened. Of these, 141 failed to meet inclusion criteria and 28 chose not to continue. The remaining 176 underwent baseline evaluation; of these 8 were excluded due to not wanting to continue (N=5) or due to MRI issues (N=3). This resulted in 168 participants who were randomized to active or sham groups.
Groups:
- Active NIR-PBM: This condition involves baseline testing, 12 weeks of Near Infrared-Photobiomodulation (NIR-PBM), and post-intervention testing. Cognitive and neuroimaging outcomes are obtained before and after the intervention. The intervention consists of a) 16 laboratory sessions of NIR-PBM given 3 times/week for 2 weeks and once weekly for 10 weeks and b) 44 home sessions of intranasal stimulation. For home sessions, participants use a standalone intranasal device on weekdays when not in the lab.
  Active NIR-PBM: Near infrared light was delivered to the head using two MedX Rehab Console systems (MedX Health, 1116). Each MedX console included a control unit and 3 superluminous light emitting diode (LED) clusters. Each LED cluster (3MedX MCT502) consisted of 52 near infrared diodes and 9 visible red diodes. The 9 red diodes were deactivated. The energy delivered by each cluster was 1 joule [J]/cm2 in 45 sec at treatment wavelength of 870 nm per each 20 min. The LED cluster has an irradiance of 22.2 mW/cm2, treats an area of 22.48 cm2, with an energy density of 26.64/cm2 per cluster (total energy of 599J/cluster). During each session, the 6 clusters were arrayed on the scalp in 2 configurations, 20 minutes per array. Each configuration targeted 6 transcranial sites, guided by the 10-20 system, for a total of 12 sites during the 40-min session. Total energy delivered was 599J/cluster X 12 sites = 7188J. Intranasal stimulation was delivered using Vielight units.
Period: Overall Study
Arm/Group | Active NIR-PBM | Sham NIR-PBM
Started | 84 | 84
Completed | 82 | 82
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active NIR-PBM | Sham NIR-PBM | Total
Number analyzed (Participants) | 84 | 84 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (4.3) | 71 (5.2) | 71 (4.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 52 | 102
  Male | 34 | 32 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 75 | 77 | 152
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 84 | 84 | 168
Education [Mean (Standard Deviation); unit: years] — Education refers to the number of years of formal education received by an individual. For example, high school graduates receive a score of 12, whereas college graduates receive score of 16. Higher scores reflect more years of education.
  years | 17 (2.3) | 16 (2.2) | 16.28 (2.24)
Montreal Cognitive Assesment [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) is a cognitive screener for dementia with scores ranging from 0 to 30. Higher scores mean better cognitive performance. For this study, participants had to score greater than the 5th percentile based on age, education, and sex-based norms (see Sachs et al. 2021).
  units on a scale | 27 (2.2) | 27 (2.0) | 27 (2.14)
Cognitive Complaints Index- Memory Scale [Mean (Standard Deviation); unit: units on a scale] — The Cognitive Complaints Index is a validated 20-item measure that assesses self-perception of cognitive change. Scores on each item range from 1 ("no change over the past 5 years") to 5 ("much worse). The first 12 items, used in this study, assess memory change and constitute the memory subscale. For the memory subscale, scores can range from 12 to 60. Participants scoring greater than 16 on the memory subscale are categorized as having subjective memory complaints. Higher scores reflect greater memory concerns.
  units on a scale | 24 (6.4) | 23 (6.3) | 23.4 (6.33)
Beck Depression Inventory-II [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory-II is a 21-item self-report scale that assesses various symptoms of depression over a two-week period. Scores range from 0 to 3 for each item, with 0 reflecting no symptoms and 3 reflecting severe concerns. Total score can range from 0 to 63. Higher scores indicate greater depression symptom severity.
  units on a scale | 6.4 (5) | 5.4 (4.7) | 5.9 (4.87)

OUTCOME MEASURES:

1. Primary Outcome: Change in Active Group ARENA Composite Score Compared to Sham Group ARENA Composite Score
Description: ARENA is a computer-based task of spatial memory-navigation that has been linked to hippocampal function and is a human analogue to the Morris water maze. ARENA consists of 9 learning trials and one final probe trial. On each learning trial, the path length and time to reach the target are recorded. On each probe trial, the percent time spent in the spatial quadrant where the target is located is recorded. The dependent variable is a total composite score consisting of mean z-scores for path length, time to reach the target, and %time in the target quadrant during the probe trial (Total Composite). Expected z-score values range from -3 to +3. A change score is computed by subtracting the baseline Total Composite z-score from the post-intervention Composite z scores. Higher scores mean better outcome.
Time Frame: Baseline; Week 12
Population: Participants included older adults with subjective cognitive complaints and a first degree relative with Alzheimer's disease. A total of 168 were randomized to active (N-84) and sham groups (N=84). The difference in N between those analyzed and enrolled relates to 4 individuals dropping out during the intervention (2 from active and 2 from sham) and 1 additional participant in the ACTIVE group who refused to complete the ARENA task.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active NIR-PBM | Sham NIR-PBM
Number analyzed (Participants) | 81 | 82
units on a scale | 0.16 (0.87) | 0.099 (0.9)
Statistical Analysis 1: Comparison: Active NIR-PBM vs Sham NIR-PBM; linear regression was used to analyze pre-post intervention changes in the active vs sham group. Covariates in regression were baseline cognitive performance, site (University of Florida, University of Arizona), age (yrs), sex (F, M) and education (years); Test type: Superiority; p = 0.573, Regression, Linear — Only 2 values, thus not necessary to adjust; The independent variable = intervention (active, sham); Covariates=baseline scores, site (Florida, Arizona), age (yrs), sex (m,f), and education (yrs)

2. Secondary Outcome: Change in Active Group Network Segregation Compared to Sham Group
Description: Functional brain network segregation (FBNS), as assessed through functional brain MRI, measures the separation between resting state connectivity networks and is indexed by Fisher Z-transformed mean correlations. FBNS is calculated as follows: Mean Within-network correlation minus Mean Between-network correlation/Mean within-network correlation. The major outcome variable was change in segregation (FBNS) from baseline to post-intervention, which has a range from -1 to +1. Larger scores indicate increased network segregation, reflecting a better outcome.
Time Frame: Baseline; Week 12
Population: Participants included 144 cognitively unimpaired healthy older individuals with a family history of AD dementia and were randomized to the active or sham intervention groups. MRI scans from 24 participants were excluded from the analyses due to scan quality control issues.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active NIR-PBM | Sham NIR-PBM
Number analyzed (Participants) | 72 | 72
units on a scale
  Default Mode Network (DMN) | 0.117 (0.42) | -0.025 (0.42)
  Frontoparietal Control Network (FPCN) | 0.090 (0.26) | 0.044 (0.26)
Statistical Analysis 1: Comparison: Active NIR-PBM vs Sham NIR-PBM; Test type: Superiority; p = 0.043, Regression, Linear — Default Mode Network Analysis: Regression was performed using permutation tests with 5000 iterations for significance and to address multiple comparisons; Covariates: Baseline network segregation values, Age, Sex, Education years, study site Baseline white matter hyperintensity volume. DOF = (1, 135)
Statistical Analysis 2: Comparison: Active NIR-PBM vs Sham NIR-PBM; Test type: Superiority; p = 0.285, Regression, Linear — Frontoparietal Control Network Analysis: Regression was performed using permutation tests with 5000 iterations for significance and to address multiple comparisons; Covariates: Baseline network segregation values, age, sex, education years, study site and baseline white matter hyperintensity volume. DOF = (1, 135)

ADVERSE EVENTS:
Time Frame: From enrollment until 3 months post intervention (approximately 6 months total).
Arm/Group | Active NIR-PBM | Sham NIR-PBM
All-Cause Mortality (participants affected / at risk) | 1/84 | 0/84
Serious Adverse Events (participants affected / at risk) | 6/84 | 5/84
Other Adverse Events (participants affected / at risk) | 15/84 | 9/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active NIR-PBM (N=84) | Sham NIR-PBM (N=84)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
chest pain (Cardiac disorders) | 1 (1) | 0 (0)
osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
dizziness and vomiting (General disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
lacrimal irritation (Eye disorders) | 1 (1) | 0 (0)
hip and back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
pulmonary embolism (Vascular disorders) | 0 (0) | 1 (2)
fainting (General disorders) | 0 (0) | 1 (1)
umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active NIR-PBM (N=84) | Sham NIR-PBM (N=84)
headache (General disorders) | 10 (12) | 6 (8)
skin cancer (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)

LIMITATIONS AND CAVEATS:
Primary limitation pertained to frequency of stimulation. For future trials, we recommend 3-4 sessions per week throughout the entire 12 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-06-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT04018092/Prot_001.pdf
  • Statistical Analysis Plan (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT04018092/SAP_002.pdf
  • Informed Consent Form (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT04018092/ICF_000.pdf